CLINICAL TRIAL: NCT00328874
Title: Mono-center, Prospective, Double-blind, Placebo-controlled, Randomized Clinical Phase IIa Trial to Assess the Safety, Tolerability, and Immediate Biological Effects of Coenzyme Q10 - nanoQuinon® in Progressive Supranuclear Palsy
Brief Title: Study About Safety and Efficacy of Coenzyme Q10 in Progressive Supranuclear Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German Parkinson Study Group (GPS) (Other)
Collaborators: MSE Pharmazeutika GmbH, Louisenstr.114D-61348 Bad Homburg, Germany (Unknown); Pitzer Stiftung (Unknown); Philipps University Marburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT: 2005-000574-40
Record Dates: First submitted 2006-05-21; First posted 2006-05-24 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2008-03

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; Coenzyme Q10
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Coenzyme Q10
- Coenzyme Q10 (Active Comparator)
  Interventions: Drug: Coenzyme Q10

INTERVENTIONS:
Drug: Coenzyme Q10

SUMMARY:
Study hypothesis:

A 6-week p.o treatment with 5 mg/Kg Coenzyme Q10 is safe and tolerable,increases the brain's metabolism and ameliorates clinical symptoms in patients with PSP.

DETAILED DESCRIPTION:
Background and Rationale:

1. Progressive Supranuclear Palsy (PSP, Steele-Richardson-Olszewski Syndrome) is a sporadic neurodegenerative disorder resulting clinically in a Parkinson syndrome (i.e. akinetic-rigid movement disorder) with prominent postural instability, oculomotor deficits, and cognitive decline (for review: Albers and Augood, 2001; Burn and Lees, 2002). With an average annual incidence of 5.3 per 100000 and an age-adjusted prevalence of 6.4 per 100000, PSP is as common as motor-neuron disease (Burn and Lees, 2002). There is no symptomatic treatment, because PSP patients do not respond to any known therapy (Albers and Augood, 2001; Burn and Lees, 2002). The progression of PSP is rapid and the median survival after onset of symptoms is 5-10 years (Albers and Augood, 2001). Presently, there is no known effective symptomatic or neuroprotective therapy for PSP.

2. Evidence suggests an impairment of mitochondrial energy metabolism in PSP (Albers and Beal, 2002):

1. Reduced cerebral glucose and ATP metabolism have been shown in functional imaging studies in PSP patients (Forster et al., 1988; Martinelli et al., 2000).
2. Cybrid cells harboring mitochondrial genes from PSP patients have decreased ATP-levels and complex I activity (Swerdlow et al., 2000; Albers et al., 2001; Chirichigno et al., 2002).
3. A tropical PSP-like tauopathy has been linked clinically and experimentally to the consumption of the fruit and teas of leaves of the tropical plant annona muricata rich in lipophilic complex I inhibitors (Caparros-Lefebvre et al., 1999; 2001). These clinical observations suggest a role for mitochondrial dysfunction in the etiology of PSP.

3.Coenzyme Q10 (CoQ10) is the physiological electron recipient of complex I. Exogenous CoQ10 (1.) enhances the electron transport by complex I and (2.) powerfully scavenges free radicals. Thus, CoQ10 has been shown to reduce the toxicity of complex I inhibitors in vitro (Menke et al., 2003) and in vivo (Beal et al., 1998

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically probable PSP (Litvan et al., 1996).
* Early stage PSP [PSP staging system ≤ III (Golbe, 1997)].
* Capability and willingness to give written informed consent to participate in the study.

Exclusion Criteria:

* Age > 85 years.
* Parkinson syndromes other than PSP (e.g. idiopathic Parkinson's disease, multiple system atrophy, diffuse Lewy body disease, FTDP17, symptomatic parkinsonism)
* Dementia [Mini Mental State Examination (MMSE) ≤ 24]
* History of epilepsy, structural brain disease, brain surgery, or electroconvulsive therapy
* History of stroke related to the onset or progression of PSP symptoms
* Arterial hypertension (systolic >180 or diastolic >110mm Hg)
* Thyroid dysfunction requiring thyroxin supplementation (CoQ10 may change its metabolism)
* Presence of other serious illnesses
* Insufficient contraception in male and pre-menopausal female participants. Accepted means of contraception are hormonal contraception, intrauterine devices, vaginal rings, preservatives, and abstinence.
* Pregnancy or lactation period
* Participation in other drug studies within 60 days before baseline visit.
* Use of CoQ10 within 60 days before baseline visit
* Use of any antioxidants (e.g. vitamin E, C) within 60 days before baseline visit
* Use of any drugs modifying mitochondrial activity within 60 days before baseline visit
* Use of statins within 60 days before baseline visit (inhibit endogenous CoQ10 production)
* Use of drugs interfering with catecholamine metabolism (e.g. reserpine, amphetamines, or monaomine oxidase-A inhibitors, methylphenidate, cinnarizine) within 30 days before baseline visit.
* Use of Levodopa within 30 days before baseline visit (CoQ10 may change its metabolism).
* An unstable dosage of CNS-active drugs (e.g. anxiolytics, hypnotics, tranquillizer, and antidepressants) within 30 days before baseline visit or throughout the study.
* An unstable dosage of other antiparkinsonian drugs within 30 days before baseline visit or throughout the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Brain Energy Metabolites measured by Magnetic Resonance Spectroscopy

SECONDARY OUTCOMES:
Slowdown of clinical progression after 6 weeks, rated with UPDRS III, PSP rating scale, PSP staging system, modified Hoehn and Yahr, FAB, MMSE, Montgomery- Asberg Depression scale, Schwab and England Score and UPDRS II
Safety and tolerability:Vital signs physical examination and safety laboratory with Blood tests and urine status.
Evaluation of occuring adverse events(AE), severe adverse events(SAE) up to 6 Weeks after the beginning of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Oertel, Professor, Principal Investigator — Neurologische Klinik der Philipps Universität Marburg
Locations (1):
- Neurologische Klinik der Philipps-Universität Marburg, Marburg, Hesse, Germany

REFERENCES:
- See also: Homepage Competence Network on Parkinson's disease sponsored by the German government, Language German, English — http://www.kompetenznetz-parkinson.de
- See also: Homepage Coordination Center for Clinical Studies to MEMSA Study, Language: German — http://www.kks-mr.de